CLINICAL TRIAL: NCT02848651
Title: A Phase II Single-Arm Study of Atezolizumab Monotherapy in Locally Advanced or Metastatic Non-Small Cell Lung Cancer: Clinical Evaluation of Novel Blood-Based Diagnostics
Brief Title: A Study of Atezolizumab as First-line Monotherapy for Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: B-F1RST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39237
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

ARMS (1):
- Atezolizumab (Experimental): Participants received 1200 milligrams (mg) of atezolizumab administered by intravenous infusion every 21 days until disease progression, loss of clinical benefit, or unacceptable toxicity (up to a total of 2 years of atezolizumab treatment).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg was administered by intravenous infusion on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit, or unacceptable toxicity (up to a total of 2 years of atezolizumab treatment).
  Other Names: MPDL3280A; RO5541267; Tecentriq

SUMMARY:
This was a Phase II, open-label, prospective, multicenter study designed to evaluate the efficacy and safety of single-agent atezolizumab as a first-line therapy in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC). In addition, the primary biomarker objective was to measure blood tumor mutational burden (bTMB) and evaluate whether it can predict for improved clinical outcome with atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed Stage IIIB-IVB NSCLC
* For participants who have received prior neo-adjuvant/adjuvant chemotherapy or chemoradiotherapy with curative intent for non-metastatic disease: a treatment-free interval of at least 6 months prior to enrollment
* Participants with any programmed death-ligand 1 (PD-L1) test result by immunohistochemistry (IHC) are eligible for the study
* Participants without a PD-L1 test result are eligible for the study
* Measurable disease per RECIST v1.1
* Adequate hematologic and end-organ function
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods among women of childbearing potential

Exclusion Criteria:

* Prior treatment with immunotherapy for any stage NSCLC, including early-stage (neoadjuvant or adjuvant) disease
* Participants with epidermal growth factor receptor (EGFR) sensitizing mutations and anaplastic lymphoma kinase (ALK) rearrangements
* Active central nervous system (CNS) metastases requiring treatment
* Spinal cord compression not definitively treated or not clinically stable
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural, pericardial effusions, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Malignancies other than NSCLC within 5 years prior to enrollment, except for those curatively treated with negligible risk of metastasis or death
* Pregnant or lactating women
* History of autoimmune disease, significant pulmonary disease, or significant cardiovascular disease
* Positive human immunodeficiency virus (HIV) or hepatitis B or C
* Active tuberculosis
* Severe infection or major surgery within 4 weeks, or oral or IV antibiotics treatment within 2 weeks prior to enrollment
* Prior treatment with or hypersensitivity to study drug or related compounds
* Prior allogeneic bone marrow or solid organ transplant
* Administration of a live, attenuated vaccine within 4 weeks prior to enrollment
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to enrollment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (20):
  - Veterans Affairs Central California Health Care System, Fresno, California
  - Memorial Regional Hospital, Hollywood, Florida
  - Florida Hospital, Orlando, Florida
  - St. Alexius Medical Center, Hoffman Estates, Illinois
  - Quincy Medical Group; Canc Ctr at Blessing Hosp, Quincy, Illinois
  - Franciscan St. Francis Health; Research Services, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Michigan Cancer Rsch Cons, Ypsilanti, Michigan
  - Virginia Piper Cancer Inst, Minneapolis, Minnesota
  - San Juan Oncology Associates, Farmington, New Mexico
  - Stony Brook University Medical Center, Stony Brook, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Levine Cancer Institute-Carolinas Medical Center; Levine Cancer Institute-Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Cancer Treatment Centers of America - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Avera Research Institute, Sioux Falls, South Dakota
  - Univ of Texas SW Medical Ctr, Dallas, Texas
  - Inova Health Care Services, Falls Church, Virginia
  - Western WA Oncology Inc PS, Lacey, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Kim ES, Velcheti V, Mekhail T, Yun C, Shagan SM, Hu S, Chae YK, Leal TA, Dowell JE, Tsai ML, Dakhil CSR, Stella P, Jin Y, Shames DS, Schleifman E, Fabrizio DA, Phan S, Socinski MA. Blood-based tumor mutational burden as a biomarker for atezolizumab in non-small cell lung cancer: the phase 2 B-F1RST trial. Nat Med. 2022 May;28(5):939-945. doi: 10.1038/s41591-022-01754-x. Epub 2022 Apr 14. PMID 35422531

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atezolizumab
Started | 153
Received Treatment | 152
Completed | 47
Not Completed | 106
Not completed — Death | 85
Not completed — Lost to Follow-up | 1
Not completed — Non-Compliance | 1
Not completed — Symptomatic Deterioration | 1
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 147
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 135
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Determined by Investigator
Description: Investigator-assessed objective response rate was defined as the proportion of participants who had a confirmed best overall response of either PR or CR per RECIST v1.1.
Time Frame: Baseline up to 32 months
Population: Efficacy and Safety analysis Population included participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Percentage of Participants | 17.1 [11.62 to 23.86]

2. Primary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 as Determined by Investigator, by Positive Versus Negative bTMB Groups
Description: Investigator-assessed PFS by RECIST v1.1 was defined as the time from the first dose of study drug to the time of PD or death from any cause during the study, whichever occurred first.
Time Frame: Baseline up to 32 months
Population: Biomarker analysis population included all participants who received at least one dose of study drug and whose tumor samples had a maximum somatic allele frequency (MSAF) >= 1%.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- bTMB Low (<16): Blood tumor mutational burdern (bTMB) Low (<16)
- bTMB High (>=16): Blood tumor mutational burden (bTMB) High (>=16)
Arm/Group | bTMB Low (<16) | bTMB High (>=16)
Number analyzed (Participants) | 91 | 28
Months | 3.55 [2.63 to 4.30] | 4.98 [1.58 to 10.81]
Statistical Analysis 1: Comparison: bTMB Low (<16) vs bTMB High (>=16); Test type: Superiority; p = 0.3502, Log Rank; Hazard Ratio (HR) = 0.80, 90% CI 2-sided [0.54 to 1.18]

3. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 as Determined by Investigator
Description: as for outcome 2
Time Frame: Baseline up to 32 months
Population: Efficacy Evaluable Population included all participants who received at least one dose of atezolizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Months | 4.14 [2.76 to 4.90]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 as Determined by Investigator
Description: Investigator-assessed DOR by RECIST v1.1 was defined as the time from initial occurrence of documented CR or PR until documented disease progression as determined by the investigator, or death, whichever occurred first.
Time Frame: Baseline up to 32 months
Population: Duration of response included a subset of participants who achieved an objective response in the efficacy evaluable population.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 26
Months | 16.33 [10.15 to NA] — Upper limit is not available because at the time of data cutoff, the upper limit of 95% CI is not estimable.

5. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 as Determined by Investigator
Description: Confirmed disease control rate (cDCR) was defined as the rate of patients with CR or PR as the best response, or SD maintained for 24 weeks, per RECIST v1.1.
Time Frame: Baseline up to 32 months
Population: Efficacy Evaluable Population included all participants who received at least one dose of atezolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Percentage | 32.9 [25.50 to 40.74]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study drug to the time of death from any cause during the study.
Time Frame: From baseline until death (up to 32 months)
Population: Efficacy Evaluable Population included all participants who received at least one dose of atezolizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Months | 14.82 [12.68 to 21.29]

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Adverse events were defined as any untoward medical occurrence in a subject administered atezolizumab, regardless of causal attribution.
Time Frame: Baseline up to 32 months
Population: Safety analyses population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 152
Percentage of Participants | 100

8. Secondary Outcome: Percentage of Participants Who Are Alive and Progression-Free (Per RECIST v1.1) at 6, 9, 12, and 18 Months by Various bTMB Quantiles
Description: A summary of the number of patients at risk and survival rate for the time points of 6, 9, 12, and 18 months.
Time Frame: Months 6, 9, 12, and 18
Population: Biomarker analysis population included all participants who received at least one dose of study drug and whose tumor samples had a maximum somatic allele frequency (MSAF) >=1%.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- bTMB <10: Blood tumor mutational burden (bTMB) <10.
- bTMB >=10: Blood tumor mutational burden (bTMb) >=10.
- bTMB <16: Blood tumor mutational burden (bTMB) <16.
- bTMB >=16: Blood tumor mutational burden (bTMB) >=16.
- bTMB <20: Blood tumor mutational burden (bTMB) <20.
- bTMB >=20: Blood tumor mutational burden (bTMB) >=20.
Arm/Group | bTMB <10 | bTMB >=10 | bTMB <16 | bTMB >=16 | bTMB <20 | bTMB >=20
Number analyzed (Participants) | 70 | 49 | 91 | 28 | 100 | 19
Percentage of Participants
  6 Months: number analyzed (Participants) | 20 | 17 | 25 | 12 | 27 | 10
  6 Months | 35.67 [23.91 to 47.43] | 34.69 [21.37 to 48.02] | 32.85 [22.85 to 42.86] | 42.86 [24.53 to 61.19] | 31.91 [22.47 to 41.34] | 52.63 [30.18 to 75.08]
  9 Months: number analyzed (Participants) | 12 | 11 | 12 | 11 | 14 | 9
  9 Months | 23.19 [12.51 to 33.86] | 22.45 [10.77 to 34.13] | 16.90 [8.60 to 25.19] | 39.29 [21.20 to 57.38] | 17.58 [9.61 to 25.55] | 47.37 [24.92 to 69.82]
  12 Months: number analyzed (Participants) | 8 | 7 | 8 | 7 | 9 | 6
  12 Months | 16.86 [6.99 to 26.74] | 14.29 [4.49 to 24.08] | 12.29 [4.79 to 19.78] | 25.00 [8.96 to 41.04] | 12.24 [5.17 to 19.31] | 31.58 [10.68 to 52.48]
  18 Months: number analyzed (Participants) | 3 | 4 | 3 | 4 | 3 | 4
  18 Months | 14.45 [4.93 to 23.98] | 8.16 [0.50 to 15.83] | 10.53 [3.36 to 17.70] | 14.29 [1.32 to 27.25] | 9.33 [2.88 to 15.78] | 21.05 [2.72 to 39.38]

9. Secondary Outcome: OS by Various bTMB Cutoff Points 16 and 20
Description: OS was defined as the time from the first dose of study drug to the time of death from any cause during the study.
Time Frame: From baseline until death (up to 32 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | bTMB <16 | bTMB >=16 | bTMB <20 | bTMB >=20
Number analyzed (Participants) | 91 | 28 | 100 | 19
Months | 13.37 [11.70 to 18.00] | 23.85 [8.77 to NA] — Upper limit is not available because at the time of data cutoff, the upper limit of 95% CI is not estimable. | 13.14 [10.48 to 17.71] | 23.85 [15.70 to NA] — Upper limit is not available because at the time of data cutoff, the upper limit of 95% CI is not estimable.
Statistical Analysis 1: Comparison: bTMB <16 vs bTMB >=16; Test type: Superiority; p = 0.1783, Log Rank; Hazard Ratio (HR) = 0.66, 90% CI 2-sided [0.40 to 1.10]
Statistical Analysis 2: Comparison: bTMB <20 vs bTMB >=20; Test type: Superiority; p = 0.0358, Log Rank; Hazard Ratio (HR) = 0.44, 90% CI 2-sided [0.23 to 0.85]

10. Secondary Outcome: Percentage of Participants With Objective Response (Per RECIST v1.1) by Various bTMB Quantiles
Description: Objective response rate was defined as the proportion of participants who had a confirmed best overall response of either PR or CR per RECIST v1.1.
Time Frame: Baseline up to 32 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- bTMB <16: Blood tumor mutational burdern (bTMB) <16.
- bTMF <20: Blood tumor mutational burden (bTMB) <20.
- bTMF >=20: Blood tumor mutational burden (bTMB) >=20.
Arm/Group | bTMB <10 | bTMB >=10 | bTMB <16 | bTMB >=16 | bTMF <20 | bTMF >=20
Number analyzed (Participants) | 70 | 49 | 91 | 28 | 100 | 19
Percentage of Participants | 7.1 [2.86 to 15.32] | 20.4 [10.51 to 33.73] | 5.5 [2.19 to 12.25] | 35.7 [19.25 to 55.54] | 6.0 [2.64 to 12.19] | 47.4 [25.17 to 69.15]
Statistical Analysis 1: Comparison: bTMB <10 vs bTMB >=10; Test type: Superiority; p = 0.0326, Cochran-Mantel-Haenszel; Differences in Rates = 13.27, 90% CI 2-sided [2.53 to 24.00]
Statistical Analysis 2: Comparison: bTMB <16 vs bTMB >=16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Rates = 30.22, 90% CI 2-sided [14.82 to 45.62]
Statistical Analysis 3: Comparison: bTMF <20 vs bTMF >=20; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Differences in Rates = 41.37, 90% CI 2-sided [22.13 to 60.61]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3 years (data cut off 26 July 2019).
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 85/152
Serious Adverse Events (participants affected / at risk) | 81/152
Other Adverse Events (participants affected / at risk) | 146/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=152)
Anaemia (Blood and lymphatic system disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 4
Septic Shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Nephritis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery occlusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=152)
Fatigue (General disorders) | 67
Oedema Peripheral (General disorders) | 21
Pyrexia (General disorders) | 12
Non-cardiac chest pain (General disorders) | 11
Chills (General disorders) | 9
Pain (General disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 41
Hypokalaemia (Metabolism and nutrition disorders) | 26
Hyponatraemia (Metabolism and nutrition disorders) | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 21
Dehydration (Metabolism and nutrition disorders) | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 17
Nausea (Gastrointestinal disorders) | 42
Diarrhoea (Gastrointestinal disorders) | 36
Constipation (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 33
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11
Weight decreased (Investigations) | 25
Blood alkaline phosphatase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 13
Alanine aminotransferase increased (Investigations) | 11
Blood creatinine increased (Investigations) | 9
Dizziness (Nervous system disorders) | 18
Headache (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 23
Depression (Psychiatric disorders) | 13
Anxiety (Psychiatric disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 14
Urinary tract infection (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 11
Pneumonia (Infections and infestations) | 9
Anaemia (Blood and lymphatic system disorders) | 24
Hypotension (Vascular disorders) | 11
Hypertension (Vascular disorders) | 10
Hypothyroidism (Endocrine disorders) | 13
Infusion related reaction (Injury, poisoning and procedural complications) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02848651/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02848651/SAP_001.pdf